CLINICAL TRIAL: NCT04329208
Title: Predictive Value of Mean Flow Velocity by TCD in Early Cerebral Vasospasm in Aneurysmal Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University 14
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral vasospasm: 13 patients developed symptomatic cerebral vasospasm detected by CT angiography and TCD
  Interventions: Device: Transcranial doppler
- Non Vasospasm: 27 patients without cerebral vasospasm
  Interventions: Device: Transcranial doppler

INTERVENTIONS:
Device: Transcranial doppler — TCD examination was performed using DWL-EZ-Dop machine Compumedics GmbH, Singen, Germany. TCD utilizes low-frequency pulsed insonation (2 MHz) to measure blood flow velocity within proximal cerebral arteries, obtaining systolic and diastolic peaks and mean flow velocities (MFV). MFV is defined as (systolic + diastolic)/3 + diastolic velocities, according to Alexandrov et al..
  Initial TCD examination was done after admission serving as a baseline state for cerebral circulation. Follow-up TCD examinations was done at fixed intervals on the first, third, fifth, seventh and tenth days of the onset of SAH.

SUMMARY:
Aim of this work is to evaluate the transcranial doppler in prediction of cerebral vasospasm in aneurysmal subarachnoid hemorrhage and also to evaluate their advantages over clinical scales in predicting CV.

DETAILED DESCRIPTION:
Cerebral vasospasm is defined as narrowing of a cerebral blood vessel enough to cause reduction in distal blood flow. Seventy percent of aSAH patients develop angiographic vasospasm but only 30% progress to develop evident neurological deficits. Cerebral vasospasm may be asymptomatic with no clinical symptoms and signs but only abnormal investigations, such as vascular stenosis by angiography or high blood flow speed by Doppler ultrasound.

Standard tests used to determine the source of bleeding and diagnose cerebral vasospasm (CV) include neuroimaging studies that administer contrast either intravenously (computed tomography angiography [CTA]) or intra-arterially (digital subtraction angiography [DSA]). Cerebral blood flow measurements using computed tomography (CT) perfusion techniques may detect the degree of cerebral ischemia in a very early stage. Although well-tolerated, these studies cannot be readily performed on the bedside and expose the patient to additional radiation, thus significantly restricting their use in daily cerebral hemodynamics monitoring. Moreover, they involve patient transportation to the CT scanner and utilization of resources such as nurses, technologists, and ancillary personnel.

Early detection of cerebral vasospasm is an important step in the way of the improvement of the outcome and the survival of aSAH patients. Transcranial duplex (TCD) is a non-invasive modality which can assess the cerebral blood vessels diameters and flow velocities that can be a useful maneuver in early detection of vasospasm after aSAH

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with spontaneous aneurysmal SAH diagnosed by non-contrast brain CT scan at the onset and confirmed by CT angiography within 72 hours of onset were included

Exclusion Criteria:

* Patient with previous history of disabling brain injuries causing focal neurological signs (e.g. motor weakness).
* Patients with poor temporal TCD window required for bedside evaluation of CV.
* Patients with decompensated systemic illness like hepatic, renal and cardiac were excluded.
* Patients with deep coma (GCS<6) were excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was a prospective study conducted on 45 consecutive aSAH patients Forty patients continued in the study and five patients were excluded because of their clinical deterioration within the first five days of the onset and or the associated decompensated systemic illness. SAH cases divided according to the presence of vasospasm into two groups; the first group included 27 cases without vasospasm, while the second group included 13 cases with vasospasm.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Mean Flow Velocity | 10 days
  TCD utilizes low-frequency pulsed insonation (2 MHz) to measure blood flow velocity within proximal cerebral arteries, obtaining systolic and diastolic peaks and mean flow velocities (MFV). MFV is defined as (systolic + diastolic)/3 + diastolic velocities.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esmael A, Belal T, Eltoukhy K. Transcranial Doppler for Early Prediction of Cognitive Impairment after Aneurysmal Subarachnoid Hemorrhage and the Associated Clinical Biomarkers. Stroke Res Treat. 2020 Nov 23;2020:8874605. doi: 10.1155/2020/8874605. eCollection 2020. PMID 33299539